CLINICAL TRIAL: NCT04122859
Title: A Randomized, Controlled, Post-market Clinical Investigation to Evaluate Zip Surgical Skin Closure Device in Comparison of Using Standard of Care Sutures for Laceration Repair in Pediatrics in an Emergency Department
Brief Title: Evaluation of Zip Device to Conventional Sutures for Laceration Repair in Pediatrics in an Emergency Department
Acronym: ZIPPED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZipLine Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Laceration of Skin
Keywords: Pediatrics

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled post-market clinical investigation that will enroll pediatric subjects requiring laceration repair. The investigation population will consist of 30 pediatric subjects fulfilling the eligibility criteria for the clinical investigation. The subjects will be randomly assigned at a 1:1 ratio to either the Zip 4 Surgical Skin Closure Device group or the Standard of Care sutures group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zip Skin Closure Device (Active Comparator): The device is a class IIa device as per Annex II of the MDD 93/42EEC, as amended by Directive 2007/47/EEC. A CE-mark was affixed in 2014. The Zip device adheres to the skin adjacent to an incision or laceration by use of pressure-sensitive skin adhesives. A combination of acrylic and hydrocolloid adhesives is used to provide a skin-friendly environment while providing the necessary tack to maintain skin adhesion during a maximum wear time of 14 days. In addition to the pressure-sensitive adhesives, the device's closure and force distribution components are made up of polyurethane monofilm, polyethylene tape, polyester and nylon.
  Interventions: Device: Zip Skin Closure Device
- Standard of Care Sutures (Active Comparator): Conventional sutures used for laceration repair
  Interventions: Device: Zip Skin Closure Device

INTERVENTIONS:
Device: Zip Skin Closure Device — The device is a CE-marked, single use, sterile medical device that is designed to provide closure speed superior to sutures, while resulting in a suture-like cosmetic outcome. It adheres to the skin adjacent to an incision or laceration by use of pressure-sensitive skin adhesives.

SUMMARY:
A prospective, randomized, controlled post-market clinical investigation that will enroll pediatric subjects requiring laceration repair. The investigation population will consist of 30 subjects fulfilling the eligibility criteria for the clinical investigation. The subjects will be randomly assigned at a 1:1 ratio to either the Zip 4 Surgical Skin Closure Device group or the Standard of Care sutures group.

DETAILED DESCRIPTION:
The commercial use of the Zip device has demonstrated applicability and acceptance in many medical specialties, including laceration closure in the Emergency Department setting. However, while clinical studies have demonstrated quantitative performance benefits of the device in orthopedic, dermatology, cardiac and cardiology specialties, no quantitative studies have been conducted in the Emergency Department setting with the device with which emergency medicine physicians may make quantitative, informed treatment choices. The Sponsor (ZipLine Medical) and the study doctor (investigator) have furthermore identified the pediatric patient population presenting for laceration repair in the Emergency Department as a group that may uniquely benefit from the use of the Zip device.

Standard care for wounds of this type require cleaning the wound, anesthetizing the wound and closing the wound with sutures that typically require subsequent removal at a later date. The Zip device is non-invasive and therefore requires no injected anesthesia or sedation for wound closure. In addition, the referenced clinical studies have demonstrated at least a 3 times speed advantage over sutures. The Zip device ease of use and consistency of outcomes enables less skilled or experienced caregivers to perform fast, efficient and excellent wound closure, which can improve department and staff efficiency, patient throughput and overall patient satisfaction. Finally, the Zip device may be removed by the patient or parent at home, eliminating a return-to-clinic visit for removal.

ZipLine Medical believes that the demonstrated benefits of the Zip device will be more pronounced with the specified pediatric population due to reduced procedure time, elimination of injected anesthesia and elimination of a return visit for suture removal. ZipLine Medical believes that this will reduce fear and anxiety in pediatric patients. Furthermore, ZipLine Medical believes that the Zip device can improve Emergency Department efficiency and patient throughput, reduce overall healthcare cost and improve overall patient (and parent) satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Between 4 to 14 years of age at the time of laceration repair.
2. Require suture closure as standard of care for simple straight wounds on trunk or extremities up to 4 cm long.
3. Low Tension Laceration, e.g. skin can be easily approximated by pinching with fingers.
4. Subject and legal representative(s) are willing and able to comply with the investigational device removal and meet the follow up visit requirements.
5. Subject and legal representative(s) have been informed of the nature, the scope and the relevance of the study.
6. Subject and legal representative(s) have voluntarily agreed to participation and have duly signed the Informed Consent Form.

Exclusion Criteria:

1. Known personal or familial history of scar hypertrophy.
2. Known or suspected allergies or hypersensitivity to non-latex skin adhesives.
3. Atrophic skin deemed clinically prone to blistering.
4. Wounds that are easily susceptible to infection as a result of exposure to unsanitary conditions ("dirty wounds").
5. Wounds that require deep dermal closure using sutures.
6. Known or suspected mental problems and/or aggressiveness that indicates that the subject might try to remove the device during the treatment period.
7. Participating in any other clinical investigation.
8. Known health condition that would affect healing in the opinion of the investigator.
9. Any subject that according to the Declaration of Helsinki is deemed unsuitable for study enrollment.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean difference in time to wound closure of the Zip 4 Surgical Skin Closure Device in comparison to conventional sutures used in a pediatric population presenting for laceration repair. | Intra operative
  These include total treatment time and duration of period starting from the preparation of procedure until protective wound dressing is applied, and including whether or not anesthesia and/or sedation was used when comparing the Zip 4 Surgical Skin Closure Device and the standard of care closure suturing

SECONDARY OUTCOMES:
Difference in Wound Evaluation Score (WES) | 10 days and 30 days post laceration repair
  A Wound Evaluation Score will be documented by an independent reviewer of photos taken at Day 0 and compared to 10 Day and 30 Day to evaluate the satisfaction and outcomes of the Zip 4 Surgical Skin Closure Device in comparison to conventional sutures used in a pediatric population presenting for laceration repair. The WES evaluates six clinical variables including incision edges, contour irregularity, width, edge inversion, inflammation and overall cosmesis. A score of 6 is considered optimal, while a score of < or =5 suboptimal.
Satisfaction of Rate of Wound Healing of Laceration Repair:satisfaction rating | 30 days post laceration repair
  Parents of patients will document the rate of wound healing satisfaction in subject post-treatment. The satisfaction rating for the Zip 4 Surgical Skin Closure Device will be compared to conventional sutures used in a pediatric population for laceration repair. The questionnaire will contain questions where the parent either will mark the most correct answer or rate on a line between 0 (Very Satisfied) to 100 (Very Dissatisfied) mm.
Pain Level for Wound Healing of Laceration Repair: visual analog scale (VAS) | Day 0 and 10 days post laceration repair
  Parents of patients will document the level of pain the patient experiences in connection to the Zip 4 Surgical Skin Closure Device and conventional sutures application and removal used in a pediatric population for laceration repair by a visual analog scale (VAS) 0 (No Pain) -100 (Worst Pain) mm
Safety by Adverse Events reported that relate to the study device | Intra operative through the end of the study at 30 days post laceration repair
  The incidence and severity of adverse events associated with the Zip 4 Surgical Skin Closure Device and Standard of Care closure sutures.

CONTACTS AND LOCATIONS:
Overall Officials: Uri Balla, MD, Principal Investigator — Kaplan Medical Center, Eehovot Israel
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT04122859/Prot_000.pdf